CLINICAL TRIAL: NCT01561014
Title: A Phase I Study of Preoperative Chemoradiation With Oxaliplatin, 5-Fluorouracil, Erlotinib and Radiation Followed by Resection and Consolidative Erlotinib for Patients With Locally Advanced Cancer of the Esophagus and Gastroesophageal Junction
Brief Title: Oxaliplatin, Fluorouracil, Erlotinib Hydrochloride, and Radiation Therapy Before Surgery and Erlotinib Hydrochloride After Surgery in Treating Patients With Locally Advanced Cancer of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007063; NCI-2009-01447 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 60106 (Other: Wake Forest University Health Sciences); NCT00499564 (obsolete NCT alias)
Record Dates: First submitted 2012-02-14; First posted 2012-03-22 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Adenocarcinoma of the Stomach; Squamous Cell Carcinoma of the Esophagus; Stage II Esophageal Cancer; Stage II Gastric Cancer; Stage III Esophageal Cancer; Stage III Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Stomach Neoplasms | interventions — Erlotinib Hydrochloride; Oxaliplatin; Fluorouracil; Radiotherapy; Radiation; Surgical Procedures, Operative; Congresses as Topic; Immunohistochemistry; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Gene Expression Profiling; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, enzyme inhibitor therapy) (Experimental): CHEMORADIOTHERAPY: Patients undergo radiation therapy QD, 5 days a week and receive fluorouracil IV continuously and erlotinib hydrochloride PO QD on days 1-38. Patients also receive oxaliplatin IV over 2 hours on days 1, 15, and 29.
  SURGERY: Within 4-8 weeks after completion of chemoradiotherapy, patients with potentially resectable disease (i.e., complete response, partial response, or stable disease) undergo surgery to remove the tumor.
  CONSOLIDATION CHEMOTHERAPY: Within 2-4 weeks after surgery, patients with tumors that demonstrate positive immunohistochemistry for EGFR and/or cyclin D1 (in the pretreatment biopsy or in the residual tumor in the esophagectomy specimen) receive consolidation chemotherapy comprising erlotinib hydrochloride PO QD for 12 weeks.
  Interventions: Drug: erlotinib hydrochloride; Drug: oxaliplatin; Drug: fluorouracil; Radiation: radiation therapy; Procedure: conventional surgery; Other: immunohistochemistry staining method; Procedure: positron emission tomography; Procedure: computed tomography; Procedure: laboratory biomarker analysis; Genetic: gene expression analysis; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: conventional surgery — Undergo surgical resection
  Other Names: surgery, conventional
Other: immunohistochemistry staining method — Correlative study
  Other Names: immunohistochemistry
Procedure: positron emission tomography — Correlative study
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Correlative study
  Other Names: tomography, computed
Procedure: laboratory biomarker analysis — Correlative study
Genetic: gene expression analysis — Correlative study
Radiation: fludeoxyglucose F 18 — Undergo F18 PET and CT scan
  Other Names: 18FDG; FDG

SUMMARY:
This phase I trial is studying the side effects and best dose of erlotinib hydrochloride when given together with oxaliplatin, fluorouracil, and radiation before surgery and alone after surgery in treating patients with locally advanced cancer of the esophagus and gastroesophageal junction. Drugs used in chemotherapy, such as oxaliplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with erlotinib hydrochloride and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving erlotinib hydrochloride after surgery may kill any tumor cells that remain after surgery

DETAILED DESCRIPTION:
OBJECTIVES:

I. The primary aim of this phase I study is to evaluate the safety of multi-drug chemotherapy (with the addition of an anti-epidermal growth factor receptor [EGFR] agent erlotinib [erlotinib hydrochloride]) and concomitant radiotherapy followed by resection and consolidative erlotinib for the treatment of locally advanced esophageal cancer as judged by the dose limiting toxicities. Correlative endpoints include an analysis of pre-treatment tumor cyclin D1 expression and EGFR expression/amplification.

III. Correlate pathologic complete response with changes in fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)-computed tomography (CT) - pre and post-chemoradiation.

OUTLINE: This is a dose escalation study of erlotinib hydrochloride

CHEMORADIOTHERAPY: Patients undergo radiation therapy once daily (QD), 5 days a week and receive fluorouracil intravenously (IV) continuously and erlotinib hydrochloride orally (PO) QD on days 1-38. Patients also receive oxaliplatin IV over 2 hours on days 1, 15, and 29.

SURGERY: Within 4-8 weeks after completion of chemoradiotherapy, patients with potentially resectable disease (i.e., complete response, partial response, or stable disease) undergo surgery to remove the tumor.

CONSOLIDATION CHEMOTHERAPY: Within 2-4 weeks after surgery, patients with tumors that demonstrate positive immunohistochemistry for EGFR and/or cyclin D1 (in the pretreatment biopsy or in the residual tumor in the esophagectomy specimen) receive consolidation chemotherapy comprising erlotinib hydrochloride PO QD for 12 weeks.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with locally advanced esophageal cancer with either squamous or adenocarcinoma histology; patients should have evidence of extension of disease into or through the wall of the esophagus (T2-4) and/or regional nodal metastasis (N1)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Non-pregnant; patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method); nursing mothers are also ineligible
* Prior treatment: Greater than one week shall have elapsed since any major surgery; no prior chemotherapy or radiotherapy is allowed
* Adequate whole blood cell (WBC) and platelets (Plt) as determined by medical oncology
* Serum creatinine =< 1.5 mg/dl
* Creatinine clearance >= 60 ml/min
* Hemoglobin (Hgb) >= 9.0 gm/dl
* Absolute neutrophil count >= 1,500/uL
* Serum total bilirubin =< 1.5 mg/dL
* Alkaline phosphatase =< 3X the upper limit of normal (ULN) for the reference lab
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than 2X ULN for the reference laboratory
* Patients must be told of the investigational nature of the study and must sign a written informed consent
* No serious medical or psychiatric illnesses which would prevent informed consent or otherwise limit survival to less than two years; no history of refractory congestive heart failure or cardiomyopathy
* Patients should be evaluated by medical oncology, radiation oncology, and surgery, and felt to by all to be suitable for trimodality therapy

Exclusion Criteria:

Patients with an active infection or with a fever >= 38.5 degrees Celsius (C) within 3 days of the first scheduled day of protocol treatment

* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current prostate surface antigen (PSA) of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry
* Patients with known hypersensitivity to any of the components of oxaliplatin
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Peripheral neuropathy >= Grade 2
* History of allogeneic transplant
* Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Toxicity rate of combination chemotherapy followed by surgery and erlotinib hydrochloride | Approximately 6 months
  Toxicity will be determined using the revised National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 3.0 for Toxicity and Adverse Event Reporting (CTCAE v3.0). The dose limiting toxicity will be defined as any of the following that can be attributal to therapy: Any grade 4 neutropenia and or any grade 4 thrombocytopenia, or any >= grade 3 non-hematologic toxicity that results in a greater than 3 day interruption of therapy.

SECONDARY OUTCOMES:
Time to progression | Approximately 4 years
Survival | Approximately 4 years
Specific characteristics that predict complete response rate (e.g., EGFR status, EGFR amplification, and cyclin D1 expression) | Over 4 years
Specific characteristics that predict complete response rate (e.g., EGFR status, EGFR amplification, and cyclin D1 expression) | Approximately 1 year
Test the predictive value of FDG-PET-CT imaging in identifying patients who will have a complete response | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Blackstock, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States